CLINICAL TRIAL: NCT02930954
Title: Combination of Gefitinib With Chemotherapy or Anti-angiogenesis as 1st Line Treatment in Advanced NSCLC Patients Detected With Bim Deletion or Low EGFR Activating Mutation Abundance
Brief Title: Gefitinib Combined With Chemotherapy or Antiangiogensis in Patients With Bim Deletion or Low EGFR Mutation Abundance
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Caicun Zhou (Other)
Responsible Party: Sponsor-Investigator, Caicun Zhou, Professor, doctor, Tongji University
Organization: Tongji University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FK1408
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Non-small-cell Lung Cancer
Keywords: NSCLC, EGFR, Bim, mutation abundance
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Pemetrexed; Gemcitabine; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Gefitinib single agent (Active Comparator): Advanced NSCLC patients with EGFR activating mutation (L858R, 19Del) received Gefitinib 250mg Qd orally until progression, intolerable toxicity or death.
  Interventions: Drug: Gefitinib
- Gefitinib combined with chemotherapy (Experimental): Gefitinib 250mg Qd combined with pemetrexed or gemcitabine plus carboplatin: Pemetrexed (500mg/m²day 1 intravenously) plus carboplatin (AUC=5,day 1,intravenously) every 21 days, Gemcitabine (1000 mg/m² days 1,d8, intravenously) plus carboplatin (AUC=5,day 1,intravenously) every 21 days
  Interventions: Drug: Gefitinib; Drug: pemetrexed or gemcitabine plus carboplatin,
- Gefitinib combined with antiangiogenesis (Experimental): Gefetinib 250mg Qd combined with bevacizumab 7.5mg/kg per 21 days
  Interventions: Drug: Gefitinib; Drug: bevacizumab

INTERVENTIONS:
Drug: Gefitinib — Patients received Gefitinib 250mg Qd orally until disease progression, intolerable toxicity or death.
  Other Names: Iressa
Drug: pemetrexed or gemcitabine plus carboplatin, — doublet chemotherapy with pemetrexed or gemcitabine plus carboplatin per 3 weeks
  Other Names: Alimita or Gimza
  Arms: Gefitinib combined with chemotherapy
Drug: bevacizumab — bevacizumab 7.5mg/kg intravenously per 3 weeks
  Arms: Gefitinib combined with antiangiogenesis

SUMMARY:
This is a single arm phase II clinical trial, which aims to evaluate the effectiveness of combination of gefitinib and doublet chemotherapy or antiangiogenesis in advanced non-small cell lung cancer patients with EGFR activating mutation, accompanied with Bim deletion or low activating EGFR mutation abundance.

DETAILED DESCRIPTION:
BIM deletion polymorphism and low EGFR mutation abundance were poor clinical response markers to EGFR-TKIs in NSCLC patients who had EGFR mutations.This is a phase II clinical trial to investigate the efficacy of combination treatment for patients harboring risk factors.

Advanced EGFR mutated NSCLC Patients with Bim deletion or EGFR low mutation abundance were randomizely divided into three treatment groups:

A:Gefitinib 250mg Qd B:Gefitinib 250mg Qd combined with doublet chemotherapy: Pemetrexed (500mg/m²day 1 intravenously) plus carboplatin (AUC=5,day 1,intravenously) every 21 days, Gemcitabine (1000 mg/m² days 1, day8, intravenously) plus carboplatin (AUC=5,day 1,intravenously) every 21 days C:Gefitinib 250mg Qd combined with bevacizumab 7.5mg/kg intravenously per 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, locally advanced or recurrent (stage IIIb and not amenable to combined modality treatment) or metastatic (stage IV) non-small cell lung cancer, anti-cancer treatment naiive
* EGFR exon 19 deletion or exon 21 L858R.
* Bim deletion by realtime PCR, or low abundance for EGFR mutation, for 19Del less than 4.9%, for L858R less than 9.5%.
* ECOG performance status of ≤ 1.
* Patients must have measurable disease according to the RECIST (version 1.1) criteria.
* Life expectancy of at least 12 weeks
* Written (signed) informed Consent to participate in the study.
* Adequate organ function as defined by the following criteria:

Liver function: SGOT (AST) and SGPT (ALT) ≤ 2.5 X ULN in the absence of liver metastases or up to 5 X ULN in case of liver metastases. Total bilirubin ≤ 1.5ULN.

Bone marrow function: Granulocyte count ≥ 1,500/mm3 and platelet count ≥100,000/mm3 and hemoglobin ≥90g/dl.

Renal function: serum creatinine ≤ 1.5 ULN or creatinine clearance ≥ 60 ml/min. (based on modified Cockcroft-Gault formula).

* For all females of childbearing potential a negative serum/urine pregnancy test must be obtained within 48 hours before enrollment. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential.

Exclusion Criteria:

* Patients with prior chemotherapy or systemic anti-cancer therapy including target therapy targeting HER family members (such as erlotinib, gefitinib, cetuximab, trastuzumab, etc). Previous adjuvant or neo-adjuvant treatment for non-metastatic disease is permitted if completed ≥ 6 months before the enrollments.
* Patients with history of any other malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer).
* Patients who have brain metastasis or spinal cord compression. It is permitted if the patient has been treated with surgery and/or radiation with evidence of stable disease for at least 4 weeks.
* Patients who are at risk (in the investigator's opinion) of transmitting human immunodeficiency virus (HIV) through blood or other body fluids.
* lactating women
* Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study.
* Unwilling to write informed consent to participate in the study or unwilling to receive follow-up
* Tumor invade big vessels or close to big vessels (less than 5mm)
* Obvious cavity or necrosis formed in the tumor, Uncontrolled hypertension, Myocardial ischemia or infarction more than stage II, cardiac insufficiency. Abnormal coagulation (INR>1.5 or PT>ULN+4, or APTT>1.5 ULN), bleeding tendency or receiving coagulation therapy
* Hemoptysis, more than 2.5ml daily
* Thrombosis in 12 months, including pulmonary thrombosis, stoke, or deep venous thrombosis.
* Unhealed bone fracture or wound for long time

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 8 weeks
  From start of anti-cancer therapy untill progression or death

SECONDARY OUTCOMES:
overall survival | 36 months
  evaluated in the 36th since treatment begain
side effect | 8 weeks
  toxicities related to anti-cancer therapy
quality of life | 24 months
  evaluated since treatment began

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD,PhD, Principal Investigator — Shanghai Pulmonary Hospital, Tongji University
Locations (1):
- Department of Oncology, Shanghai pulmonary hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Share the patient characteristics, results of test, treatment and outcome.